CLINICAL TRIAL: NCT06156683
Title: Kesimpta (Ofatumumab) Pregnancy and Infant Safety Study Using Real World Data
Brief Title: Kesimpta Pregnancy and Infant Safety Study Using Real World Data
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157G2405; EUPAS106133 (Other: ENCePP)
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Kesimpta; ofatumumab; real world data
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Kesimpta-exposed: exposure to Kesimpta during the risk period
  Interventions: Other: Multiple sclerosis disease modifying drug
- MSDMD-exposed: exposure to at least one Multiple sclerosis disease modifying drug (MSDMD) (other than Kesimpta) during the risk period
  Interventions: Other: Multiple sclerosis disease modifying drug
- MSDMD-unexposed: no exposure to Kesimpta or any other Multiple sclerosis disease modifying drug (MSDMD) during the risk period
  Interventions: Other: Multiple sclerosis disease modifying drug

INTERVENTIONS:
Other: Multiple sclerosis disease modifying drug — There is no treatment allocation. Women with multiple sclerosis with a recorded pregnancy outcome during the inclusion period will be recruited.

SUMMARY:
The study is an observational retrospective cohort study using longitudinal secondary data. Pregnant women with MS are assessed for exposure to Kesimpta and other MS disease modifying drugs (MSDMD) and followed up for adverse pregnancy and infant outcomes.

DETAILED DESCRIPTION:
Outcomes among Kesimpta exposed pregnancies are compared primarily to MSDMD-exposed pregnancies and secondarily to MSDMD-unexposed pregnancies.

The main research question is to determine whether the exposure during pregnancy to Kesimpta increases the risk of adverse pregnancy and infant outcomes in women with MS.

The risk period is defined as the 1st trimester of pregnancy for analyses of Major congenital malformations and the entire duration of pregnancy for all other outcomes.

The data for this study is retrieved from data sources from Denmark, Sweden, and the US, based on an assessment of feasibility.

ELIGIBILITY:
Inclusion Criteria:

The following overall criteria for study inclusion are applied:

* Pregnancy with a recorded start and end of pregnancy outcome (live birth, spontaneous abortion, elective termination, stillbirth, or ectopic pregnancy) during the inclusion period
* Age 18-49 years at index date
* A diagnosis of MS before the index date. This inclusion criterion is based on diagnosis codes, as recorded in the different data sources
* Availability of information on exposure to MSDMDs and maternal baseline characteristics for a minimum of 12 months before the index date

In addition, the following outcome and objective specific inclusion criteria are applied:

* For analyses of MCMs in live births (primary objective): pregnancy ending in at least one live birth
* For analyses of spontaneous abortion, elective termination of pregnancy, stillbirth, preeclampsia, eclampsia (secondary objectives): pregnancy ending in at least one live birth, spontaneous abortion, elective termination, stillbirth, or ectopic pregnancy
* For analyses of preterm birth, SGA (secondary objectives): pregnancy ending in at least one live birth
* For analyses of MCMs among live births, spontaneous abortions, stillbirths, and elective terminations (exploratory objective): pregnancy ending in at least one live birth, spontaneous abortion, still birth, or elective termination
* For analyses of neonatal infection: live newborn
* For analyses of SII: newborn alive at 29 days after birth

Exclusion Criteria:

The following overall criteria for exclusion are applied:

* Pregnancy exposed to a MSDMD that have a known teratogenic effect, determined based on the date of prescription, estimated supply duration, and the drug-specific window of clearance
* Pregnancy exposed to a non-MSDMD that have a known moderate to high teratogenic effect, determined based on the date of prescription, estimated supply duration, and the drug-specific window of clearance

The following outcome specific exclusion criteria are applied:

* For analyses of MCMs and exploratory analyses of MCMs: pregnancies with a record of a chromosomal abnormality or a genetic syndrome
* For analyses of preterm birth, pre-eclampsia, eclampsia and SGA, pregnancies involving multiples
* For Kesimpta and MSDMD-exposed cohorts: pregnancies not exposed during the outcome specific risk period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The overall study population consists of women with MS with a recorded pregnancy outcome during the inclusion period. Pregnancies exposed to MSDMDs with a known teratogenic effect or non-MSDMDs with a known moderate to high teratogenic effect are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of major congenital malformations (MCM) among live births | First year of life, up to 12 months
  The primary outcome of interest concerns MCMs occurring in pregnancies ending in at least one live birth. MCMs are defined as defects that have either cosmetic or functional significance to the child (e.g., a cleft lip)

SECONDARY OUTCOMES:
Number of participants with spontaneous abortions | Up to 9 months
  Also termed miscarriage, is defined as the unintended loss of an intrauterine pregnancy less than 20 weeks of gestation (<20 weeks).
Number of participants with elective termination of pregnancy | Up to 9 months
  Defined as the intentional termination of pregnancy at any time in gestation for any reason. When possible, reasons for elective termination are captured and classified as elective termination of pregnancy for fetal anomaly or for other reasons.
Number of participants with stillbirths | Up to 9 months
  Defined as the unintended fetal death occurring at or after 20 weeks of gestation.
Number of participants with preterm births | Up to 9 months
  Defined as live births less than 37 weeks of gestation (<37 weeks). Elective caesarean deliveries or inductions prior to 37 completed weeks will be described separately.
Number of participants with preeclampsia | Up to 9 months
  Preeclampsia is defined as the new-onset of hypertension with a systolic blood pressure greater than or equal to 140 mmHg and/or diastolic blood pressure greater than or equal to 90 mmHg at or after 20 weeks of gestation with proteinuria and/or endorgan dysfunction (renal dysfunction, liver dysfunction, central nervous system disturbances, pulmonary edema, and thrombocytopenia).
Number of participants with eclampsia | Up to 9 months
  Eclampsia is defined as the new onset of generalized tonic-clonic seizures in a woman with preeclampsia
Number of participants small for gestational age (SGA) | Up to 9 months
  Defined as a birth weight lower than the 10th percentile for gestational age and sex using the national standards in each study country in a live birth

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No